CLINICAL TRIAL: NCT01560988
Title: Treatment of Bronchial Asthma With Borage and Echium Seed Oils
Brief Title: Borage and Echium Seed Oils for Asthma
Acronym: Borage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Wake Forest University (Other)
Responsible Party: Principal Investigator, Joshua Boyce, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2010p002041
Record Dates: First submitted 2012-03-09; First posted 2012-03-22 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Asthma
Keywords: Asthma; Borage; Echium; Botanical
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Borage and Echium Seed Oils (Experimental): Borage and echium oil capsules administered daily for six weeks, then a 6 week washout period, followed by ingestion of placebo (corn oil capsules) daily for 6 weeks.
  Interventions: Drug: Borage and Echium Seed Oils; Dietary Supplement: Corn oil pills
- Corn oil pills (Experimental): Corn oil capsules daily for six weeks, then a 6 week washout period, followed by ingestion of Borage and echium oil capsules daily for 6 weeks.
  Interventions: Drug: Borage and Echium Seed Oils; Dietary Supplement: Corn oil pills

INTERVENTIONS:
Drug: Borage and Echium Seed Oils — 4.0 g/day borage seed oil and 7.0 g/day echium seed oil. Pills will be taken three times per day for six weeks.
Dietary Supplement: Corn oil pills — Corn oils pills will be taken three times per day for six weeks.

SUMMARY:
This study plans to look at whether borage and echium seed oils (natural oils from two plants) help decrease asthma symptoms and affect cells involved in inflammation. The investigators also want to look at how these plant oils decrease the generation of inflammatory cells in people with asthma.

DETAILED DESCRIPTION:
To evaluate the mechanisms by which borage seed oil and echium seed oil block mediator generation in asthma, we performed a cross-over trial design to reduce the numbers of patients needed for the study. Each treatment period was six weeks with a six-week washout period. For simplicity all power calculations are made assuming a single factor or predictor variable and a single result or outcome variable. We focused on changes in mediator generation by effector cells. Calculations below suggest that we have resolution to pick up clinically meaningful effects of potentially important explanatory variables with acceptable or high power.

1. Study Design The goals were to examine the mechanisms that underlie the effects of borage seed oil and echium seed oil on proinflammatory mediator production by effector leukocytes.

In the treatment arm, subjects consumed 4.0 g/day borage seed oil and 7.0 g/day echium seed oil (containing totals of ~1.6 g/day of GLA and ~0.9 g/day of SDA). The oils were packaged in capsules each of which contained 1 gram of oil. Therefore subjects will ingest 10 capsules a day (3 in the morning, 3 in the afternoon, and 4 in the evening) with meals. In the placebo arm, subjects took matching capsules containing corn oil; three 1 gram capsules in the morning and afternoon, and four in the evening, with meals.

The study began with a screening visit. All subjects had physician-diagnosed asthma. All performed a baseline set of lung function measurements. They entered a 2-week run-in period during which they kept a diary of peak flows, asthma symptoms, and beta agonist use. Subjects were instructed in peak flow technique and asked to perform three maneuvers each time. The maneuver was considered technically sufficient if the variation in the values obtained on the three attempts are with 10% of each other, and the highest value was recorded in a diary. Subjects whose diaries were > 80% complete entered the study and were randomly assigned to active treatment or placebo. Spirometry was repeated. Blood was taken for fatty acid composition of plasma and leukocytes, LT generation, and DNA for genotyping at the LTC4S locus. Subjects were provided with peak flow diaries, instructed in the appropriate performance or peak flow maneuvers, and asked to record morning and evening peak flow each day (reflecting the best of three efforts each time). After three weeks of treatment, diary cards will be collected and spirometry repeated. After six weeks of treatment, blood was drawn for safety monitoring, for measurements of fatty acids in plasma and leukocytes, and for the functional analyses. Spirometry was repeated. Subjects then entered a six-week washout period. Two weeks before the end of this period they again started to keep diary cards. At the conclusion of the 6-week washout period they entered the cross-over treatment phase (six weeks) which followed the same protocol as the first treatment period with assessment of fatty acid analyses, cellular function studies, safety monitoring, and spirometry. Pregnancy testing was performed before and after each treatment period. Dairy cards (with peak flow monitoring results) will be collected at each visit (3 week intervals during the placebo and active treatment arms of the study).

3. Statistical Analyses

a. Power Calculations - For simplicity all power calculations are made assuming a single factor or predictor variable and a single result or outcome variable. While a number of correlated outcomes will be investigated, we will focus on changes in mediator generation and levels of enzyme expression. Calculations below suggest that we have resolution to pick up clinically meaningful effects of potentially important explanatory variables with acceptable or high power.

i. Biochemical Endpoints - Power is based on paired t-tests comparing continuous measures of response between treatment and placebo. We assume 40 subjects will be available after allowing for a drop out rate of 20% from our original sample of 50 subjects. For the endpoint of leukotriene production by leukocytes, the power calculations suggested that we will have 80% power to detect a true within-subject difference of 0.8 of the within-subject SD between treatment and placebo with an α value of 0/05. On the basis of our previous studies, we assume a within-subject coefficient of variation (CV) of 13% for LTC4 generation. This will translate to an approximate detectable difference from 10.5% in these parameters.Using a paired two-sided t-test and prior mean(standard deviation) estimates for the placebo of .001464 ( .002268) and for the borage oil of .000289( .000709) , we would need 40subjects for 80-90% power at a 0.05 level of significance to detect a change in LTC4S transcript, protein, and enzymatic activity of 50% between placebo and borage arms.

b. Analysis Plan - Initially, we will present descriptive statistics (mean, standard deviation, range) for all endpoints to treatment and placebo groups. We will also present graphical plots of all measures across the study and for each group within each period. For the 2x2 crossover study, we will compare the treatment and control on each endpoint separately by employing a generalized mixed model approach with the predictors: group(sequence), patient nested within group as a random effect, period(dichotomous), treatment(dichotomous), and seasonality(dichotomous), with unstructured covariance. We will utilize mixed model diagnostics such as residual plots to assess goodness of fit.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years to 65 years of age
2. Stable physician diagnosed asthma with FEV1 of greater than 50% of predicted but less than 90% of predicted or less than 90% of known best and an asthma control questionnaire(ACQ) < 1.5.

Exclusion Criteria:

1. Pregnant or nursing
2. Smoking history of > 10 pack years or active smoking within the past year.
3. Due to possible effects on LT biosynthesis, use of the following asthma treatments within the preceding month will be exclusion criteria:

   * LT modifying drugs (zileuton, montelukast, zafirlukast)
   * theophylline
   * oral steroids
   * dietary supplements with fatty acids or other products that may interfere with LT generation.
4. Treatment within the previous three months with omalizumab (monoclonal antibody directed against IgE)
5. Subjects will not be permitted to take non-steroidal anti-inflammatory drugs in the week prior to any measurements of ex vivo LT generation because of their effects on LT biosynthesis via inhibition of prostaglandin generation.
6. A history of aspirin-sensitive asthma will be an exclusion criterion as the effects of GLA/SDA on prostanoid biosynthesis have not been adequately elucidated.
7. Significant abnormalities in CBC, differential white cell count, renal function, and liver function, or urinalysis.
8. No subjects will have any serious co-morbid medical condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Boyce, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Asthma Research Center Website — http://asthmabwh.org

RESULTS

PARTICIPANT FLOW:
Groups:
- First Borage and Echium, Then Corn Oil: Borage and Echium Seed Oils: 4.0 g/day borage seed oil and 7.0 g/day echium seed oil. Pills will be taken three times per day for six weeks, followed by a 6 week washout. Then, subjects were crossed over to receive corn oil (10 g) daily for six weeks
- First Corn Oil, Then Borage and Echium Seed Oil: Corn oil pills will be taken for six weeks, followed by a 6 week washout. Then subjects received borage and echium oil tablets for six week.
Period: First Intervention (Six Weeks)
Arm/Group | First Borage and Echium, Then Corn Oil | First Corn Oil, Then Borage and Echium Seed Oil
Started | 32 | 30
Completed | 22 | 26
Not Completed | 10 | 4
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 3 | 0
Period: Washout (Six Weeks)
Arm/Group | First Borage and Echium, Then Corn Oil | First Corn Oil, Then Borage and Echium Seed Oil
Started | 22 | 26
Completed | 20 | 24
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2
Period: Second Intervention (Six Weeks)
Arm/Group | First Borage and Echium, Then Corn Oil | First Corn Oil, Then Borage and Echium Seed Oil
Started | 20 | 24
Completed | 18 | 22
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Population: Patients with physician diagnosed asthma between 18 and 65 years of age
Groups:
- All Study Participants: Participants were randomized to receive either borage and echium oils first, and corn oil second, or vice versa
Arm/Group | All Study Participants
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 62
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 19
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: Cellular Changes That Occur With Borage and Echium Seed Oil Supplementation
Description: Primary outcome measures will be changes in the generation of LTC4 production by granulocytes. This was calculated by the difference between the amount produced at the start of each arm and at the end of each arm (i.e., two values were obtained in each arm and used to calculate the difference, and the differences were compared as a delta-delta).
Time Frame: Assessed at 2, 8, 14, and 20 weeks
Population: We analyzed all samples available, including from subjects who did not complete the entire protocol (i.e., 40 subjects crossed over and completed both arms, but 44 completed the corn oil and 44 completed the borage and echium arm, and the overlap was incomplete). Thus, the number of subjects differs from the total number of subjects per arm.
Measure: Mean (Standard Deviation); unit: ng
Groups:
- Borage and Echium Seed Oils: Borage and echium seed oils will be taken for six weeks.
  Borage and Echium Seed Oils: 4.0 g/day borage seed oil and 7.0 g/day echium seed oil. Pills will be taken three times per day for six weeks.
- Corn Oil Pills: Corn oil pills will be taken for six weeks.
  Corn oil pills: Corn oils pills will be taken three times per day for six weeks.
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 39 | 38
ng | 5.06 (15.7) | 2.56 (15.0)

2. Primary Outcome: Change in LTB4 Production
Description: Primary outcome measures will be changes in the generation of LTB4 production by granulocytes. This was calculated by the difference between the amount produced at the start of each arm and at the end of each arm (i.e., two values were obtained in each arm and used to calculate the difference, and the differences were compared as a delta-delta). A negative number implies that the level of LTB4 produced by granulocytes at the end of the arm was less than the amount produced at the start of the arm, while a positive number means that more was generated at the end than at the beginning.
Time Frame: At 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Groups:
- Corn Oil Pills: Corn oil pills will be taken for six weeks.
  Corn oil pills will be taken three times per day for six weeks.
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 39 | 38
ng | -.99 (8.73) | 0.12 (6.21)

3. Secondary Outcome: Measure of DHA in Cell Pellets
Description: Secondary outcome measures include changes in concentrations of omega 3 fatty acids in cell pellets, indicating incorporation of botanical oil metabolites in cell membrane lipids.. This was calculated by the difference between the amount present at the start of each arm and at the end of each arm (i.e., two values were obtained in each arm and used to calculate the difference, and the differences were compared as a delta-delta).
Time Frame: Assessed at 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 39 | 39
ng | 1.18 (8.51) | -1.01 (11.00)

4. Secondary Outcome: Lung Function
Description: Changes in lung function (forced expiratory volume in 1 second) will be assessed via spirometry at each visit. This was calculated by the difference between the FEV1 at weeks 2 and 8 versus weeks 14 and 20. The differences were compared as a delta-delta. A negative number for this parameter means that the FEV1 was lower at the end of the arm than at the beginning, while a positive number means that the FEV1 was higher at the end.
Time Frame: Assessed at 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- Borage and Echium Seed Oils: Borage and echium seed oils will be taken for six weeks.
  Borage and Echium Seed Oils: 4.0 g/day borage seed oil and 7.0 g/day echium seed oil.
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 42 | 39
Percent change | -.12 (6.7) | 0.22 (5.77)

5. Secondary Outcome: Plasma Level of Gamma Linolenic Acid (GLA)
Description: Changes in plasma level of gamma linolenic acid (GLA), a major constituent of Borage oil, as a measure of compliance. This was calculated by the difference between the amount produced at the start of each arm and at the end of each arm (i.e., two values were obtained in each arm and used to calculate the difference, and the differences were compared as a delta-delta).
Time Frame: Measurements obtained at 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 39 | 39
ng | 6.11 (10.2) | -.25 (2.32)

6. Secondary Outcome: Number of Subjects Bearing a Polymorphic Variant of LTC4 Synthase
Description: All individuals will be genotyped at the LTC4S locus.
Time Frame: two weeks
Population: We analyzed all samples available including those who did not complete both arms of the protocol. Therefore the number of subjects in the two arms are not identical.
Measure: Number; unit: participants
Groups:
- All Study Participants: All study participants, regardless of arm assignment, were genotyped at the LTC4S locus.
Arm/Group | All Study Participants
Number analyzed (Participants) | 42
participants | 10

7. Secondary Outcome: Asthma Control
Description: Changes in asthma control will be assessed via the Asthma Control Questionnaire (ACQ) at each visit. The ACQ is a 6-point questionnaire that reflects the degree of asthma activity. Each point is assigned a scale of 0-5, with 5 being the worst. Thus, the range is from 0 (no asthma symptoms) to 30 (severe asthma symptoms). For each arm, we generate two values (week 2 vs. week 8 and week 14 vs.week 20). These values are then averaged for each arm to obtain the final single value. A negative number implies improved symptoms.
Time Frame: Assessed at 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Change in ACQ points
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 42 | 39
Change in ACQ points | -.18 (0.64) | -.12 (.50)

8. Secondary Outcome: Measure of EPA in Cell Pellets
Description: as for outcome 3
Time Frame: Assessed at 2, 8, 14, and 20 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 37 | 37
ng | .094 (2.01) | -0.02 (2.10)

9. Secondary Outcome: Change in Activity of LTC4 Synthase
Description: Differences in LTC4S activity while receiving borage/echium oils versus corn oil stratified by LTC4S genotype. We analyzed the genotype for 32 subjects for the borage arm and 30 subjects for the placebo arm.
Time Frame: Days 0, 42, 84, and 126
Population: Since this is a crossover study, 30 of 32 who completed the borage arm also completed the corn oil arm. The data presented reflect the effects of borage/echium versus corn oil for individuals with two wild type alleles (AA) versus those with one variant allele (CC or AC).
Measure: Mean (Standard Deviation); unit: ng/million cells
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 42 | 39
ng/million cells
  Genotype AA: number analyzed (Participants) | 32 | 30
  Genotype AA | .95 (11.3) | -.10 (7.83)
  Genotype AC or CC: number analyzed (Participants) | 10 | 9
  Genotype AC or CC | 18.0 (18.5) | 11.7 (25.9)

10. Secondary Outcome: Genotype-specific Differences in Change in Lung Function While Receiving Borage and Echium Oils Versus Corn Oil.
Description: FEV1 was measured in all subjects at the beginning and end of both study arms. Subjects were genotyped at LTC4S locus and those bearing at least one A to C polymorphism were compared with those bearing two A alleles.
Time Frame: 0, 42, 84, and 126 days
Population: We analyzed all samples available including subjects who did not complete the entire protocol. Therefore the number of subjects analyzed differs from the total number of subjects per arm.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
Number analyzed (Participants) | 42 | 39
Liters
  Genotype AA: number analyzed (Participants) | 32 | 29
  Genotype AA | -.02 (.23) | -.02 (.16)
  Genotype AC or CC: number analyzed (Participants) | 10 | 9
  Genotype AC or CC | 0.08 (.25) | .18 (.22)

ADVERSE EVENTS:
Time Frame: The study ran for 20 weeks and data were collected over that time frame.
Arm/Group | Borage and Echium Seed Oils | Corn Oil Pills
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/38
Other Adverse Events (participants affected / at risk) | 14/42 | 6/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Borage and Echium Seed Oils (N=42) | Corn Oil Pills (N=38)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma deterioration (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — Increased use of rescue inhaler or decreased lung function
Gastrointestinal distress (Gastrointestinal disorders) | 6 (6) | 2 (2) — Constipation, gassiness, heatburt
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Elevated liver enzymes (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes